CLINICAL TRIAL: NCT01375673
Title: Effects of Exercise Training on Fluid Instability in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRI 09-228
Record Dates: First submitted 2010-10-08; First posted 2011-06-17 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure
Keywords: Exercise; Heart Failure; Mixed Effects Modeling
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Exercise: Walking Strength Training Bicycling
  Interventions: Other: Exercise
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Other: Exercise — Walking Strength Training Bicycling
  Arms: Exercise

SUMMARY:
Heart Failure (HF) is a significant healthcare concern in the US, with a 120% rise in mortality rates over 15 years costing the country an estimated $37.2 billion in 2009. Veterans are currently impacted at a rate of 5.2%, and cost an average of $14,959/individual/year for those utilizing the VA's Healthcare services. Research has shown that exercise training (ET) improves aerobic capacity, endothelial dysfunction, quality of life, and the ability to tolerate activity within the overall HF population. The purpose of this study is to examine the effects of structured exercise training and specific types of exercise training, walking, bicycling, and resistance training, on the symptom of fluid volume over load or edema in advanced heart failure patients.

DETAILED DESCRIPTION:
Background: Heart Failure (HF) is a significant healthcare concern in the US, with a 120% rise in mortality rates over 15 years costing the country an estimated $37.2 billion in 2009. Veterans are currently impacted at a rate of 5.2%, and cost an average of $14,959/individual/year for those utilizing the VA's Healthcare services. Research has shown that exercise training (ET) improves aerobic capacity, endothelial dysfunction, quality of life, and the ability to tolerate activity within the overall HF population. Animal models have emerged to explain some of the underlying mechanisms for the pathologic expression of symptoms and the links to ET. A translational link has not yet been explored between the animal models and human symptom expression.

Objectives: The long-term goal of this research program is to develop an exercise training (ET) program that effectively decreases fluid shift variability in HF patients, while being safely implemented in the home environment and remotely monitored by a healthcare provider within a nurse-lead HF Clinic. The purpose of the proposed research project is to determine if ET alters fluid status of patients with HF as compared to those under standard treatment of care. The central hypothesis is that a combined weight-bearing aerobic and resistance ET protocol will reduce (stabilize) 24-hour weight and bioelectrical impedance patterns of variability, as evaluated via mixed-effects regression modeling, greater than any other form of ET protocol.

Methods: Design: Using established experimental design techniques implemented in an innovative manner, a between-group design is used within the experimental arm employing a single subject, multiple-baseline design. The use of such technique allows for the subjects to be their own controls, while also allowing for statistical between group comparisons.

Subjects and Setting: 60 subjects meeting inclusion/exclusion criteria will be enrolled from the VA HF Clinic and outpatient VA cardiology clinics within 50 miles of Columbia, South Carolina. Subjects will be randomized to the exercise or usual care groups.

Procedures: The exercise protocol lasts 12 weeks, with subjects being randomized to order of ET. Weight-bearing aerobic ET will be walking on a treadmill; non-weight-bearing aerobic ET will be stationary bicycling; and resistance ET will be lower body isolation ET. Fluid stability is the concept of day-to-day variability of movement of intra-cellular fluid to extra-cellular space. Fluid stability will be assessed using 24-hour weight and bioelectrical impedance and quantified statistically using mixed effect modeling.

Data Analysis: Statistical analysis will utilize a longitudinal mixed-effects regression model, modeling variability over time for the subjects individually, as well as within groups. Additionally, main effects (time and group) and interaction effects (time by group) will be assessed.

Status: Funding began September 1, 2010. The study was transferred to Dorn VAMC in Columbia, SC in March of 2011. Currently the study is in the final phase of data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Heart Failure
* Ability to Walk
* Over 21

Exclusion Criteria:

* Renal Failure
* Inability to walk
* Physician exclusion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Boyd, PhD, Principal Investigator — Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC
Locations (1):
- Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 98 subjects were screened. Of the 98, 15 were female, 21 meet both inclusion and exclusion criteria, and 16 began the enrollment process. Of those 16 subjects, 1 died prior to full consent, 1 choose not to enroll.
Groups:
- Standard of Care: Standard of care
Period: Overall Study
Arm/Group | Exercise | Standard of Care
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Standard of Care | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Ejection Fraction [Count of Participants; unit: Participants] — those at or below 25% Ejection Fraction, those 26-40% and those greater than 41% per Echocardiogram.
  Participants
    25% and less EF | 3 | 3 | 6
    26-40% EF | 2 | 3 | 5
    41% and greater EF | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Bioelectrical Impedance Change
Description: The extracellular fluid was calculated and reported to demonstrate Fluid Instability. A Bioelectrical Impedance Monitor was utilized to attain these measures.
Time Frame: baseline, week 16, week 24
Population: BioImpedence/Extracellular vs intracellular fluid analyzed daily for 24 weeks. Daily values compressed into mean for week x 24 weeks.
Measure: Mean (Standard Deviation); unit: Percentage of Extra Cellular Fluid
Arm/Group | Exercise | Standard of Care
Number analyzed (Participants) | 7 | 7
Percentage of Extra Cellular Fluid
  Baseline-Week 4 | 47.52 (1.5) | 47.1 (1.35)
  Intervention-Week 16 | 41.27 (2) | 46.8 (1.45)
  Maintenance-Week 24 | 42.1 (1.7) | 47.0 (1.4)

2. Secondary Outcome: Body Weight Change
Description: Body weight was assessed via a home weight scale. Patients recorded their morning body weight in pounds up to 1 decimal point. The daily values were then used to create a weekly standard deviation to represent variability of daily weight. The standard deviation was then meaned for phase of the study. The values reported represent absolute weight means across participants.
Time Frame: baseline, week 16, week 24
Population: Daily weight was recorded in pounds and then converted into a weekly standard deviation
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Exercise | Standard of Care
Number analyzed (Participants) | 7 | 7
Pounds
  Baselline-Weeks 1-4 | 249 (2.14) | 256 (1.88)
  Intervention-Weeks 5-16 | 242 (0.45) | 260 (1.9)
  Maintenance-Weeks 17-24 | 258 (0.95) | 261 (1.85)

3. Secondary Outcome: Health Outcome Measures Change
Description: Health Outcomes were measured with a Daily Heart Failure Symptom Questionnaire. The likert scale was converted to a continuous scale ranging from 0-15 for each of the 10 questions. The higher scores are more indicative of active HF symptoms while lower scores are lack of active HF symptoms. Range for this total score is 0-150.
Time Frame: baseline, week 16, week 24
Population: The Heart Failure Questionnaire was assessed as a daily measure with weekly mean and SD being reported for each phase. The Likert Scale was converted to a continuous scale from 0 to 15 cm and scores added together for the 10 questions to get a total score.
Measure: Mean (Standard Deviation); unit: Total Points
Arm/Group | Exercise | Standard of Care
Number analyzed (Participants) | 7 | 7
Total Points
  Baseline-Week 4 | 25.05 (1.48) | 27.25 (1.52)
  Intervention-Week 16 | 18.2 (1.7) | 28.25 (1.75)
  Maintenance-Week 24 | 28.55 (3) | 29.5 (1.8)

ADVERSE EVENTS:
Time Frame: 2 years
Description: No difference in definition
Arm/Group | Exercise | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Limited patient population due to the clinic, strict limitations of inclusion/exclusion criteria and the distance many participants would have had to travel to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes